CLINICAL TRIAL: NCT06247852
Title: Persistent Pain After Cesarean Delivery - A Danish Multicenter Cohort Study
Status: Completed | Type: Observational
Sponsor: Nordsjaellands Hospital (Other)
Responsible Party: Principal Investigator, Patricia Duch, Consultant, MD, Nordsjaellands Hospital
Other Study IDs: 101
Record Dates: First submitted 2024-01-08; First posted 2024-02-08 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Cesarean Section Complications; Cesarean Section; Cesarean Delivery; Persistent Pain; Chronic Pain; SMS; Questionnaire
Keywords: persistent pain; chronic pain; Danish cohort; cesarean section; cesarean delivery; acute on chronic pain; post operative pain; SMS questionnaire
MeSH Terms: conditions — Chronic Pain; Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In Denmark, around 12,700 patients undergo Cesarean delivery (CD) annually, constituting approximately 20% of all childbirths in the country. Worldwide, the number is increasing each year, with more than 20 million CD performed annually.

Postoperative pain after CD is typically moderate to severe in intensity and still constitutes a significant challenge, balancing effective pain relief and potential side effects. Correlations between moderate to severe acute pain and the development of persistent pain after CD is still unclear.

Postsurgical persistent pain is a significant, often unrecognized clinical problem that causes distress and diminishes the quality of life for patients. Despite advances in understanding the factors contributing to persistent postsurgical pain and an increased focus on identifying patients at risk, the management and prevention of postsurgical persistent pain are still inadequate.

It is important to gain further insights into this population, and we have a unique opportunity to do so by following the national cohort from the ongoing Danish multicenter cohort study on pain after cesarean section (ClinicalTrials.gov Identifier: NCT06012747) over an extended follow-up period.

This involves continued prospective registration of Patient-Reported Outcome Measures (PROM) collected by SMS-based questionnaires in the months and years after the CD, thereby investigating the occurrence of both acute and persistent pain after CD.

The outcomes are focused on pain levels, the impact of pain on physical function and neuropathic pain characteristics in the months and years following the CD. The study also aims to explore the relationship between persistent and acute pain.

DETAILED DESCRIPTION:
The Study Protocol is attached in full-text (Study Documents).

ELIGIBILITY:
Inclusion Criteria:

* Patients who, after participating in the Danish multicenter cohort study on pain after cesarean delivery (ClinicalTrials.gov Identifier: NCT06012747), consent to continue to receive questionnaires about persistent pain.
* Planned cesarean delivery in spinal anesthesia
* Patients who speak and read Danish
* Patients with a smartphone that can receive an SMS with a link to a questionnaire that can be opened online.

Exclusion Criteria:

• <18 years of age

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients having a cesarean section
Study Population: Patients, aged > 18 years, who undergo planned cesarean delivery under spinal anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 477 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-06-10 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Persistent pain | after 6 months
  The percentage of patients reporting pain equivalent to an NRS score > 3 after 6 months

SECONDARY OUTCOMES:
Severe pain during the last 24 hours. | Assessments are conducted at 5 weeks, 2, 3, 6, and 12 months, and after that every 6 months until 3 years after surgery.
  NRS 0-10
Severe pain at rest during the last 24 hours. | Assessments are conducted at 5 weeks, 2, 3, 6, and 12 months, and after that every 6 months until 3 years after surgery.
  NRS 0-10
Use of analgesic medication in the past week due to pain (Paracetamol, Non-Steroidal Anti-Inflammatory Drug, opioid). | Assessments are conducted at 5 weeks, 2, 3, 6, and 12 months, and after that every 6 months until 3 years after surgery.
  Yes/No
Pain's affect on daily activities | Assessments are conducted at 5 weeks, 2, 3, 6, and 12 months, and after that every 6 months until 3 years after surgery.
  1-5: Not at all, a little, to some extent, to a great extent, cannot do due to pain.
Pain's affect on engaging in strenuous physical activity. | Assessments are conducted at 5 weeks, 2, 3, 6, and 12 months, and after that every 6 months until 3 years after surgery.
  1-6: Not at all, a little, to some extent, to a great extent, cannot do due to pain, I don't know - I haven't tried.
Pain's affect on meeting the infant's needs. | Assessments are conducted at 5 weeks, 2, 3, 6, and 12 months, and after that every 6 months until 3 years after surgery.
  1-5: Not at all, a little, to some extent, to a great extent, cannot do due to pain.
Pain's affect on sleep. | Assessments are conducted at 5 weeks, 2, 3, 6, and 12 months, and after that every 6 months until 3 years after surgery.
  1-4: Not at all, a little, to some extent, to a great extent.
Pain's affect on mood. | Assessments are conducted at 5 weeks, 2, 3, 6, and 12 months, and after that every 6 months until 3 years after surgery.
  1-4: Not at all, a little, to some extent, to a great extent.
Pain/discomfort when sitting down or standing up from a chair. | Assessments are conducted at 5 weeks, 2, 3, 6, and 12 months, and after that every 6 months until 3 years after surgery.
  1-5: Not at all, a little, to some extent, to a great extent, cannot do due to pain.
Pain/discomfort when walking on stairs. | Assessments are conducted at 5 weeks, 2, 3, 6, and 12 months, and after that every 6 months until 3 years after surgery.
  1-5: Not at all, a little, to some extent, to a great extent, cannot do due to pain.
Pain/discomfort when getting in or out of bed. | Assessments are conducted at 5 weeks, 2, 3, 6, and 12 months, and after that every 6 months until 3 years after surgery.
  1-5: Not at all, a little, to some extent, to a great extent, cannot do due to pain.
Pain/discomfort when carrying the infant. | Assessments are conducted at 5 weeks, 2, 3, 6, and 12 months, and after that every 6 months until 3 years after surgery.
  1-5: Not at all, a little, to some extent, to a great extent, cannot do due to pain.
Pain/discomfort when sitting up for less than 30 minutes. | Assessments are conducted at 5 weeks, 2, 3, 6, and 12 months, and after that every 6 months until 3 years after surgery.
  1-5: Not at all, a little, to some extent, to a great extent, cannot do due to pain.
Pain/discomfort if sitting up for more than 30 minutes. | Assessments are conducted at 5 weeks, 2, 3, 6, and 12 months, and after that every 6 months until 3 years after surgery.
  1-6: Not at all, a little, to some extent, to a great extent, cannot do due to pain, I don't know - I haven't tried.
Pain/discomfort when moving around at home. | Assessments are conducted at 5 weeks, 2, 3, 6, and 12 months, and after that every 6 months until 3 years after surgery.
  1-5: Not at all, a little, to some extent, to a great extent, cannot do due to pain.
Pain/discomfort if walking for more than 30 minutes. | Assessments are conducted at 5 weeks, 2, 3, 6, and 12 months, and after that every 6 months until 3 years after surgery.
  1-6: Not at all, a little, to some extent, to a great extent, cannot do due to pain, I don't know - I haven't tried.
Pain/discomfort when bending down. | Assessments are conducted at 5 weeks, 2, 3, 6, and 12 months, and after that every 6 months until 3 years after surgery.
  1-5: Not at all, a little, to some extent, to a great extent, cannot do due to pain.
Pain/discomfort during or after sexual intercourse. | Assessments are conducted at 5 weeks, 2, 3, 6, and 12 months, and after that every 6 months until 3 years after surgery.
  1-7: Not at all, a little, to some extent, to a great extent, cannot do due to pain, I don't know - I haven't tried, I prefer not to answer.
Pins and needles, tingling or stabbing sensations in or around the area of the surgery? | Assessments are conducted at 5 weeks, 2, 3, 6, and 12 months, and after that every 6 months until 3 years after surgery.
  Yes/No
Electric shock like sensation or jabbing feelings in the skin area in or around the area of the surgery? | Assessments are conducted at 5 weeks, 2, 3, 6, and 12 months, and after that every 6 months until 3 years after surgery.
  Yes/No
Heat or burning sensations in or around the area of the surgery? | Assessments are conducted at 5 weeks, 2, 3, 6, and 12 months, and after that every 6 months until 3 years after surgery.
  Yes/No
Pain caused by the lightest of touches in or around the area of the surgery? | Assessments are conducted at 5 weeks, 2, 3, 6, and 12 months, and after that every 6 months until 3 years after surgery.
  Yes/No
Pain caused by cold temperatures in or around the area of surgery? | Assessments are conducted at 5 weeks, 2, 3, 6, and 12 months, and after that every 6 months until 3 years after surgery.
  Yes/No

OTHER OUTCOMES:
Recall of acute pain at 12 and 24 hours after CD | Asked 12 months after CD.
  Exploratory
Percentage of patients experiencing pain with an NRS > 3 | 1, 2, 3, and 12 months, as well as 1,5; 2; 2,5 and 3 years after cesarean delivery.
  Exploratory
Association between severe acute pain (NRS > 6) during the first 24 hours and the occurrence of persistent pain at 6 and 12 months after CD. | 12 months
  Exploratory
Prevalence of chronic pain before pregnancy. | 6 months
  Exploratory
Prevalence of chronic pain before pregnancy and its association with the development of persistent pain | 1, 2, 3, and 12 months, as well as 1,5; 2; 2,5 and 3 years after cesarean delivery.
  Exploratory
6. Association between uterine exteriorization versus in situ repair in CD and the occurrence of persistent pain | 1, 2, 3, and 12 months, as well as 1,5; 2; 2,5 and 3 years after cesarean delivery.
  Exploratory

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Duch, MD, Principal Investigator — University Hospital of Copenhagen, Hillerød, Denmark; Helene Nedergaard, MD, Ph.D, Study Director — University Hospital of Southern Denmark, Kolding; Christoffer Jørgensen, Dr. Med., Study Director — University Hospital of Copenhagen, Hillerød, Denmark; Kim Wildgaard, MD, Ph.d., Study Chair — University Hospital of Copenhagen, Herlev, Denmark
Locations (1):
- Department of Anesthesiology, Copenhagen University Hospital, North Zealand Hillerød, Hillerød, Denmark

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2024-01-30): https://cdn.clinicaltrials.gov/large-docs/52/NCT06247852/Prot_000.pdf